CLINICAL TRIAL: NCT01810406
Title: A Randomized Controlled Trial of Epidural Volume Extension During a Combined Spinal-Epidural Technique for Labor Analgesia.
Brief Title: Epidural Volume Extension During a Combined Spinal-Epidural Technique for Labor Analgesia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Ronald George, Principal Investigator, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IWK - 1013037
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Pregnancy; Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epidural Volume Extension (Experimental): CSE with 10 ml EVE
  Interventions: Procedure: CSE with 10 ml EVE
- No Epidural Volume Extension (Active Comparator): CSE without EVE
  Interventions: Procedure: CSE without EVE

INTERVENTIONS:
Procedure: CSE with 10 ml EVE — Combined Spinal-Epidural (CSE) with 10 ml Epidural Volume Extension (EVE)
  Other Names: Normal Saline
  Arms: Epidural Volume Extension
Procedure: CSE without EVE — Combined Spinal-Epidural (CSE) without Epidural Volume Extension (EVE)
  Arms: No Epidural Volume Extension

SUMMARY:
Combined spinal-epidurals (CSE) involve the injection of pain relief medication into the cerebral spinal fluid (CSF) and the insertion of an epidural catheter in the epidural space to continue to give pain relief medication. During a CSE, after injection of the medication in the CSF and before inserting the epidural catheter, if normal saline is injected into the epidural space, there may be an increase in pain relief and an increase in the level of numbness. This injection of saline in the epidural space to increase pain relief and numbness is termed epidural volume extension (EVE). The purpose of this study is to determine if there is a benefit for EVE to improve labor analgesia (pain relief) using CSE in pregnant laboring patients.

DETAILED DESCRIPTION:
Regional analgesia (pain relief) for labor can be an epidural, a spinal or a combination of the two. Combined spinal-epidurals (CSE) are popular because of their rapid pain relief and high patient satisfaction. At the IWK Health Centre, many anesthesiologists routinely use this method of pain relief. It involves the injection of pain relief medication into the cerebral spinal fluid (CSF) and the insertion of an epidural catheter (slim plastic tube) in the epidural space to continue to give pain relief medication. The epidural space is located just outside the CSF. In order to insert the epidural catheter, some anesthesiologists inject 2-4 ml of saline in the epidural space to help the catheter go in. During a CSE, after injection of the medication in the CSF and before inserting the epidural catheter, if normal saline is injected into the epidural space, there may be an increase in pain relief and an increase in the level of numbness. This injection of saline in the epidural space to increase pain relief and numbness is termed epidural volume extension (EVE).

Thus far, studies on EVE have all been done in patients undergoing surgery with spinal anesthesia and not solely for analgesia. The purpose of this study is to determine if there is a benefit for EVE to improve labor analgesia (pain relief) using CSE. We will study 60 women requesting labor pain relief. Half these women will receive a CSE without EVE, which is the present standard of care. The other half will receive a CSE with 10 ml of saline for EVE before inserting the epidural catheter. We will then determine if there is a benefit for EVE by observing for a difference between the two groups with respect to the level of numbness, the amount and speed of pain relief and the intensity of leg weakness. We hypothesize that injecting 10 ml of saline for EVE using CSE may improve the amount and speed of pain relief while decreasing side effects such as leg weakness. If there were a benefit to EVE, this would be a simple and inexpensive method for improving pain relief in laboring women.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous parturients requesting regional analgesia for labour pain with singleton, vertex presentation fetuses at 37-42 week gestation in active labor with cervical dilation < 5 cm.
* American Society of Anesthesia physical status class I & II (ASA I - Healthy, ASA II - mild and controlled systemic disease, e.g. controlled essential hypertension)
* Age ≥ 18 years (Standard within the obstetrical anesthesia literature)
* English-speaking

Exclusion Criteria:

* Contraindications to neuraxial analgesia (i.e. coagulopathy, systemic infection, neuropathy)
* Conditions associated with abnormal spinal anatomy which can affect local anesthetic spread (i.e. scoliosis, spina bifida, spinal instrumentation)
* Conditions associated with an increased risk of a cesarean delivery (i.e., history of uterine anomaly or surgery, morbid obesity (Body Mass Index ≥ 35 kg/m2)
* Clinically significant diseases of pregnancy such as pregnancy-induced hypertension or preeclampsia (defined as systolic blood pressure (SBP) > 160mmHg, diastolic blood pressure (DBP) > 110mmHg and/or requiring antihypertensive treatment or associated with significant proteinuria)
* Severe maternal cardiac disease
* Known fetal anomalies /intrauterine fetal demise
* Patient enrollment in another study involving a study medication within 30 days
* Any other physical or psychiatric condition which may impair their ability to cooperate with study data collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Sensory dermatome level | 30 minutes
  As determined by non-traumatic pinprick test

SECONDARY OUTCOMES:
Analgesia | 30 minutes
  As assessed by numeric rating scale (NRS)
Motor block | 30 minutes
  Assessed using a modified Bromage scale

OTHER OUTCOMES:
Side effects | 30 minutes
  Includes hypotension, pruritus, nausea, fetal distress, and local anesthetic toxicity related side effects
Additional analgesia given | 30 minutes
  Either self-administered by the patient via PCEA (Patient Controlled Epidural Analgesia) button, or administered by an anesthesiologist

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Zaphiratos, MSc MD FRCPC, Principal Investigator — IWK Health Centre; Ronald B George, MD FRCPC, Principal Investigator — IWK Health Centre
Locations (1):
- Women's and Obstetric Anesthesia, IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Zaphiratos V, George RB, Macaulay B, Bolleddula P, McKeen DM. Epidural Volume Extension During Combined Spinal-Epidural Labor Analgesia Does Not Increase Sensory Block. Anesth Analg. 2016 Sep;123(3):684-9. doi: 10.1213/ANE.0000000000001281. PMID 27088994